CLINICAL TRIAL: NCT07384286
Title: Behavioral Reinforcement Intervention for Greater Health Trajectories After Childhood Cancer (BRIGHT)
Acronym: BRIGHT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 286561
Record Dates: First submitted 2026-01-15; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Survivors of Childhood Cancer
Keywords: Lifestyle; Survivors of childhood cancer

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial with waitlist design and crossover of control group, plus a parallel group randomized controlled trial for effectiveness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Register-based follow-up (No Intervention): Participants in NOPHO-CARE Sweden who are randomized to not being contacted regarding BRIGHT but will only undergo register-based follow-up within NOPHO-CARE Sweden
- Waitlist control with cross-over (Active Comparator): Active participation in BRIGHT. Randomized to waitlist control and start of intervention after 6 months.
  Interventions: Behavioral: Lifestyle Management
- Immediate intervention (Experimental): Active participation in BRIGHT and randomized to immediate start of the intervention.
  Interventions: Behavioral: Lifestyle Management

INTERVENTIONS:
Behavioral: Lifestyle Management — Person-centered lifestyle support
  Arms: Immediate intervention; Waitlist control with cross-over

SUMMARY:
Survivors of childhood cancer have a substantially increased risk of long-term health problems in adulthood, including cardiovascular disease, metabolic disorders, psychological morbidity, and impaired health-related quality of life (HRQoL). These risks are partly related to cancer treatment exposures but are also strongly influenced by modifiable lifestyle factors such as physical activity, diet, body weight, and cardiometabolic risk factors. Although healthy lifestyle behaviors are known to reduce morbidity and mortality in this population, many adult childhood cancer survivors do not meet current lifestyle recommendations and rarely receive structured, tailored support to change health behaviors.

The Behavioral Reinforcement Intervention for Greater Health Trajectories (BRIGHT) study aims to evaluate whether a person-centered, remotely delivered lifestyle intervention can improve health-related quality of life and key health markers in adult survivors of childhood cancer with an unhealthy lifestyle. The intervention focuses on increasing physical activity and improving dietary habits through structured video-based coaching delivered by trained health promoters over a 26-week period.

BRIGHT is conducted within NOPHO-CARE Sweden, a national population-based cohort of childhood cancer survivors, and uses a register-based randomized controlled design with two randomization steps. First, eligible participants are randomized to be offered the intervention or not, enabling evaluation of the population-level effect of offering the intervention through long-term register-based follow-up. Second, participants who consent to active participation are randomized to immediate or delayed start of the intervention, allowing controlled assessment of short-term intervention effects.

The primary research question is whether the BRIGHT lifestyle intervention leads to a clinically meaningful improvement in health-related quality of life, measured by the PROPr utility index derived from PROMIS-29, compared with a control period. Secondary questions address whether the intervention improves physical activity, cardiorespiratory fitness, muscle strength, diet quality, body weight, blood pressure, and cardiometabolic and biological markers, including epigenetic age acceleration. The study also examines feasibility, adherence, and scalability of delivering a person-centered lifestyle intervention within a national survivorship follow-up structure.

In addition, BRIGHT investigates whether offering the intervention to the full eligible population leads to long-term reductions in cardiovascular disease, metabolic disease, psychiatric morbidity, and mortality, using national health registers. By combining individual-level efficacy and population-level effectiveness within a single study framework, BRIGHT aims to generate robust evidence to inform future preventive care and long-term follow-up strategies for adult survivors of childhood cancer.

DETAILED DESCRIPTION:
Survival after childhood cancer has improved substantially, resulting in a growing population of adults exposed to cancer treatment early in life. Adult survivors of childhood cancer are at markedly increased risk of long-term adverse health outcomes, including cardiovascular disease, cardiometabolic disorders, psychological morbidity, and reduced health-related quality of life (HRQoL). While treatment-related factors contribute to these risks, modifiable lifestyle behaviors-particularly physical activity, diet, and body weight-play a central role in shaping long-term health trajectories. Evidence indicates that healthy lifestyle behaviors may yield even greater absolute risk reduction in childhood cancer survivors than in the general population. However, many survivors do not meet recommended lifestyle guidelines and are rarely offered structured, tailored, and sustained behavioral support within routine follow-up care.

The Behavioral Reinforcement Intervention for Greater Health Trajectories (BRIGHT) study is designed to evaluate a person-centered, remotely delivered lifestyle intervention targeting physical activity and dietary habits in adult survivors of childhood cancer with an unhealthy lifestyle. The study is embedded within NOPHO-CARE Sweden, a national population-based survivorship cohort that integrates registry data, patient-reported outcomes, and biological samples. This infrastructure enables both short-term evaluation of intervention efficacy and long-term assessment of population-level effectiveness using national health registers.

Study Design Overview BRIGHT is a pragmatic, register-based randomized controlled trial employing a two-step randomization design to simultaneously address efficacy and real-world effectiveness. The first randomization occurs at the population level within NOPHO-CARE Sweden, where eligible individuals are randomized to be offered the intervention or not. This allows evaluation of the long-term health impact of offering a lifestyle intervention at scale, independent of individual uptake, using register-based follow-up.

The second randomization occurs among participants who consent to active participation in the intervention and study-specific assessments. These participants are randomized to immediate or delayed (waitlist) start of the intervention. This design enables controlled comparisons of short-term intervention effects while ensuring that all actively participating individuals eventually receive the intervention.

Study Population The study targets adult (≥18 years) survivors of childhood cancer who are participants in NOPHO-CARE Sweden and report an unhealthy lifestyle, defined as insufficient physical activity and/or overweight or obesity. Individuals with established cardiovascular disease or other medical conditions that would make participation unsafe are excluded from active participation. Eligibility is determined using existing cohort data and baseline assessments.

Intervention The BRIGHT intervention consists of a structured, person-centered lifestyle coaching program delivered entirely through video-based sessions. Participants engage in 16 scheduled sessions over a 26-week period with trained health promoters who have expertise in behavioral science and lifestyle change. Sessions are conducted weekly during the initial phase of the intervention and biweekly thereafter.

The intervention focuses on supporting participants to increase physical activity and improve dietary habits in line with international recommendations. Using a person-centered approach, participants and health promoters collaboratively identify individualized goals, barriers, and facilitators, and regularly review progress. The intervention emphasizes sustainable behavior change rather than short-term performance targets and is tailored to each participant's preferences, capacities, and life circumstances. The intervention does not include pharmacological treatment or medical decision-making and does not replace or modify routine healthcare.

Data Collection and Assessments Study-specific assessments are conducted remotely and primarily in participants' home environments, with guidance and oversight provided via video visits by research nurses. Assessments are performed at baseline, at follow-up points aligned with intervention timing, and at longer-term follow-up for trajectory analyses.

Data collection integrates:

* Patient-reported outcomes, including health-related quality of life and lifestyle behaviors;
* Objective measurements of physical activity, fitness, body composition, and blood pressure;
* Functional performance tests conducted under video supervision;
* Self-collected capillary blood samples for laboratory analyses of cardiometabolic and biological markers.

All methods used are validated, low-risk, and suitable for remote administration. Standardized protocols and quality control procedures are applied to ensure data reliability.

Outcomes and Follow-up The primary objective of BRIGHT is to determine whether participation in the lifestyle intervention results in a clinically meaningful improvement in health-related quality of life compared with a control period. Secondary objectives address changes in physical activity, fitness, diet, cardiometabolic risk factors, and biological markers, as well as sustainability of effects over time.

Beyond individual-level outcomes, BRIGHT evaluates the long-term effectiveness of offering the intervention at the population level. Participants randomized in the first step are followed longitudinally through national health registers to assess incidence of cardiovascular disease, metabolic disease, psychiatric morbidity, healthcare utilization, and mortality. This approach enables evaluation of whether implementing a lifestyle intervention within a national survivorship follow-up structure translates into meaningful reductions in long-term disease burden.

Feasibility and Scalability An additional objective of BRIGHT is to assess feasibility, adherence, and scalability of delivering a person-centered lifestyle intervention within a national cohort. Metrics such as uptake, retention, adherence to intervention sessions, and completion of assessments are examined to inform future implementation. By embedding the trial within NOPHO-CARE Sweden, BRIGHT evaluates delivery under real-world conditions rather than in a highly selected research setting.

Safety and Ethical Considerations BRIGHT is designed as a minimal-risk behavioral intervention. Physical assessments are conducted under professional supervision via video, with predefined safety criteria and procedures for managing abnormal findings. Participants with clinically concerning measurements are advised to seek routine medical care, but no clinical treatment decisions are made within the study.

All data are pseudonymized and stored in secure research environments in accordance with national and European data protection regulations. Analyses are conducted within protected systems that prevent export of individual-level data. Results are reported only in aggregate form.

Significance BRIGHT is the first national register-based randomized controlled trial in Sweden to evaluate a fully remote, person-centered lifestyle intervention in adult survivors of childhood cancer. By combining individual-level efficacy evaluation with population-level effectiveness assessment, the study aims to generate robust evidence to inform preventive strategies and long-term follow-up care. If successful, BRIGHT may provide a scalable model for integrating structured lifestyle support into survivorship care for childhood cancer survivors at the national level.

ELIGIBILITY:
Inclusion Criteria:

* Participant in NOPHO-CARE Sweden
* Performing <150 min moderate-vigorous physical activity per week and/or body mass index 28-35.

Exclusion Criteria:

* Pre-existing diagnosis of heart failure or coronary artery disease
* Uncontrolled hypertension, defined as >180/100 mmHg
* Other medical reasons that the intervention or outcome assessments are considered unsafe (as decided by a study physician)
* Inability to perform the intervention or outcome assessments due to lack of mobile device (computer, tablet or telephone) with internet access or language barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | from Baseline until 6 months
  The primary outcome will be change in HRQoL using the PROPr utility index, derived from patient-reported outcome measures information system (PROMIS)-29.

SECONDARY OUTCOMES:
Physical activity | From baseline until six months for comparison between groups and until 18 months for trajectories.
  Physical activity will be measured by triaxial accelerometers (Axivity, model AX3).
Cardiorespiratory fitness | From baseline until six months for comparison between groups and until 18 months for trajectories.
  Cardiorespiratory fitness will be estimated using the 2-minute step test
Handgrip strength | From baseline until six months for comparison between groups and until 18 months for trajectories.
  Grip strength will be measured with the Jamar Plus+ dynamometer
Lower limb strength | Change from baseline until six months for comparison between groups and until 18 months for trajectories.
  Lower limb strength will be tested with the Chair Rise-5 repetitions
Diet | Change from baseline until six months for comparison between groups and until 18 months for trajectories.
  Riksmaten Flex questionnaire
Body mass index | From baseline until six months for comparison between groups and until 18 months for trajectories.
  Body weight will be assessed with a provided digital Seca 807 scale. Weight will be assessed after voiding, during a video meeting with a research nurse. The research nurse will ensure participants use the scale on a hard surface and follow standardized weighing procedures to minimize measurement variability. Body height will be taken from clinical information from outpatient clinic visits, registered in the Swedish Childhood Cancer Registry.
Blood pressure | Change from baseline until six months for comparison between groups and until 18 months for trajectories.
  Blood pressure will be done according to best practices for home-based blood pressure monitoring.
Patient-reported outcome measures | Change from baseline until six months for comparison between groups and until 18 months for trajectories.
  Patient-reported outcomes of fatigue, sleep, and pain, reported with PROMIS-29.
Glucose metabolism | Change from baseline until six months for comparison between groups and until 18 months for trajectories.
  Assessed with HbA1c from dried blood spots.
Lipid metabolism | Change from baseline until six months for comparison between groups and until 18 months for trajectories.
  Total cholesterol, HDL, LDL, triglycerides, and apolipoproteins from dried blood spots.
Metabolic profiles of diet intake | Change from baseline until six months for comparison between groups and until 18 months for trajectories.
  Untargeted metabolomics from dried blood spots will be analyzed.
Epigenetic age acceleration | Change from baseline until six months for comparison between groups and until 18 months for trajectories.
  Epigenetic age acceleration will be assessed from epigenetic clocks from DNA extracted from dried blood spots.
Cardiometabolic, cardiovascular, and psychiatric morbidity | From end of intervention until 2, 5, and 10 years.
  Will be assessed from register-based follow-up of randomization 1.
Mortality | From end of intervention until 5 and 10 years.
  From register-based follow-up of randomization 1.
Health economics | Until 5 years after randomization 1.
  Health economic evaluation of the intervention, using information from EQ-5D-5L and actual healthcare costs from register-based follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum för livsstilsintervention, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet.